CLINICAL TRIAL: NCT01059045
Title: Prospective Controlled Study Evaluating Cryocontact Therapy of Infantile Hemangiomas of Preterm Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitement was much slower than anticipated.
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Rangmar Goelz, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CryoHaem
Record Dates: First submitted 2010-01-28; First posted 2010-01-29 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2004-08

CONDITIONS: Hemangioma of Preterm Infants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cryocontact therapy (Experimental)
  Interventions: Procedure: cryocontact therapy
- Control (No Intervention)
  Interventions: Procedure: cryocontact therapy; Other: Control

INTERVENTIONS:
Procedure: cryocontact therapy — cryocontact therapy of hemangioma is realized by using liquid nitrogen cooled metal devices
Other: Control — No intervention
  Arms: Control

SUMMARY:
Prospective controlled study evaluating cryocontact therapy of infantile hemangiomas of preterm infants

Principal investigator: Rangmar Goelz, MD Coworkers: M Möhrle, M Moll, HM Häfner, W Schippert, C Meisner, M Röcken, CF Poets

Background Despite their frequent occurrence, there is no established therapeutic procedure for localized infantile hemangioma in preterm infants. A PubMed search with the key words hemangioma, controlled study, infant or childhood revealed five studies (1-5), none of them included preterm infants, even though low birth weight and prematurity have been described as the most significant risk factors

Aim:

To evaluate cryocontact therapy of infantile hemangioma (IH) of 1 - 10 mm diameter in preterm infants <=34 weeks of gestational age (GA) using a liquid nitrogen cooled metal at the Department of Neonatology at the Tuebingen University Hospital.

Method:

In a prospective controlled study, preterm infants <= 34 weeks GA with at least 2 IH should be randomized to have one treated with cryocontact therapy using a liquid nitrogen cooled metal (-196°C), while the other one is left untreated. Primary endpoint is an intact skin at the site of the hemangioma at 1 year corrected age . The study starts at August 1st, 2004. Cryocontact is done by 3 trained dermatologist (MM, HMH, WS), outcome documentation, including photodocumentation, by 2 neonatologist (RG, MoMo).

Statistical Analysis: A sample size of 25 intrapersonal pairs of treated and untreated IH is needed to show a significant difference with alpha=0.05 and beta=0.9 between treated IH and controls, assuming that 5% of the treated IH and 40% of the controls have an unsuccessful primary outcome. Documentation will be made on standardized forms and the data will be transferred to Excel. Biometric calculations will be handled with SAS 9.1.3. for Windows using Fisher´s Exact Test for difference in proportions.

Ethics:

The study is approved by the Ethics Committee of Tuebingen University Hospital; all parents must give written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants <=34 weeks GA with hemangioma

Exclusion Criteria:

* no hemangioma

Ages: 1 Day to 11 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2004-08; Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Hemangioma outcome | 1 year
  skin status

CONTACTS AND LOCATIONS:
Overall Officials: Rangmar Goelz, MD, Principal Investigator — University Hospital